CLINICAL TRIAL: NCT01341041
Title: Wound Irrigation: Comparison of Normal Saline With Chlorous Acid Chlorine Dioxide Solution
Brief Title: Chlorine Dioxide Versus Saline for Wound Irrigation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Jonathan Valente MD, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0334-03
Record Dates: First submitted 2011-04-11; First posted 2011-04-25 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Wound - in Medical Care
MeSH Terms: interventions — chlorine dioxide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- chlorine dioxide (Experimental): 2 arms
  Interventions: Biological: chlorine dioxide
- saline (Active Comparator): one time wash with 50-100cc of normal saline
  Interventions: Biological: saline

INTERVENTIONS:
Biological: chlorine dioxide — one time wash with 50ppm CD solution
  Arms: chlorine dioxide
Biological: saline — one time wash with 50-100 cc normal saline
  Arms: saline

SUMMARY:
This research is being done because the investigators are trying to examine the safety and effectiveness of this wound cleaning liquid, CACD (chlorine dioxide). The investigators are trying to see if this liquid has the ability to decrease infection rates and decrease the scarring effects from the healing process. In animal studies, CACD has been shown to decrease scar formation and decrease the risk of wound infections. CACD is also used for the treatment of burns to decrease infection rates and improve wound healing. CACD is not FDA approved for this specific use, but it is FDA and USDA approved for reducing bacterial contamination on meat and food products for human consumption. In addition, an investigational drug (IND) application has been submitted to the FDA for this study. The FDA has approved the use of this solution for this study.

ELIGIBILITY:
Inclusion Criteria:

* 18-100 years old
* simple laceration requiring irrigation & sutures
* patient has method of contact
* patient is willing to return to ED in 3-4 mths

Exclusion Criteria:

* immunocompromised
* consult required for repair
* diabetic
* require antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2004-08; Primary Completion 2007-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
cosmesis | 72 hrs post-ED visit
  Cosmesis will be assessed by taking pictures of the wound at presentation, upon receiving sutures, 48-72 hrs later, and 3-4 mths later. At 3-4 mths the patient will rate how well they think the wound healed, via a visual analog scale. At that time, two blinded ER physicians will do this as well. They will also designate a wound evaulation score, based on criteria that will be provided to them. Two blinded plastic surgeons will assess all photographs, visual analog scores. and wound evaluation scores, and provide their own visual analog scale assessment of how well each wound healed.

CONTACTS AND LOCATIONS:
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States